CLINICAL TRIAL: NCT03536793
Title: Study of Tumour Regulatory Molecules as Markers of Malignancy in Pancreatic Cystic Lesions
Brief Title: Tumour Regulatory Molecules in Early Pancreatic Cancer Detection
Acronym: TEM-PAC
Status: Recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Other Study IDs: R2224
Record Dates: First submitted 2018-04-25; First posted 2018-05-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cancer of Pancreas; Pancreas Cyst
Keywords: Early detection of pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pancreatic cysts: Samples (urine, serum, whole blood and cystic fluid) will be taken from 50 patients with pancreatic cysts on follow-up. These will be sent to the University of Hull for analysis of tumour regulatory molecules (e.g. TF, AM). Some of the cystic fluid and the whole blood sample will either be analysed at the University of Hull or a commercial laboratory for proteomic and genomic data. Collection will occur on the same day of the participants' routinely indicated procedure.
- Pancreatic cancers: Samples (urine and serum) will be taken from 50 patients diagnosed with pancreatic cancer (resectable and non-resectable). These will be sent to the University of Hull for analysis of tumour regulatory molecules (e.g. TF, AM).
- Benign hepatopancreatobiliary conditions: Samples (urine and serum) will be taken from 80 age- and gender-matched control patients - 20 patients with acute pancreatitis and a non-resolving pseudocyst, 20 undergoing cholecystectomy for stones, 20 undergoing cholecystectomy for inflammation and 20 patients undergoing investigations for dyspepsia (normal control subgroup). These will be sent to the University of Hull for analysis of tumour regulatory molecules (e.g. TF, AM).

SUMMARY:
The effective diagnosis of pancreatic cancer is often quite challenging, due to a lack of disease-specific symptoms, resulting in the majority of patients presenting with advanced disease, with an associated dismal prognosis. Earlier detection of pancreatic cancer, at a stage where surgery is feasible, would greatly increase the 5-year survival rate. Detecting pancreatic cancer early is therefore vital to improve the prognosis for these patients.

Pre-cancerous pancreatic cysts are an early indicator of malignant transformation. The ideal screening test would be capable of detecting pancreatic cancer at these initial stages. Current procedures for pancreatic cancer diagnosis are invasive, uncomfortable and costly, and can be considered unnecessary in those cysts found to be benign.

We propose to study a number of tumour regulatory molecules that have been the subject of research in laboratories at the University of Hull (e.g., tissue factor (TF), adrenomedullin (AM) using enzyme-linked immunosorbent assays (ELISA) tests) that have been studied in the context of carcinogenic transformation in more common malignancies but have yet to be fully tested in pancreatic malignant transformation. The recent introduction of platform technologies at the University of Hull has broadened this area of investigation by giving us access to next generation genomic sequencing and proteomic analyses of small amounts of tissue samples. We intend to analyse pancreatic cystic fluid samples using these technologies to discover new regulatory molecules.

Altogether, his study will measure the levels of novel regulatory molecules and genetic changes involved with pancreatic cancer carcinogenesis using a combination of conventional techniques (e.g. ELISA) and state-of-the-art platform technologies in pancreatic cysts from those patients in whom cancer may be suspected, to determine the potential of these molecules to serve as markers to detect early changes towards pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

General

* Capable of giving written informed consent
* Age ≥18 years

Pancreatic Cancer Cohort

- Diagnosed with localised pancreatic cancer amenable to resection (distal pancreatectomy, total pancreatectomy or Whipple's procedure).

OR - Diagnosed with inoperable localised pancreatic cancer and referred for further management (malignant control subgroup).

Pancreatic Cysts Cohort

- Presence of cystic lesions where MDT have agreed further diagnostic intervention procedures (including FNA/EUS) necessary.

OR - Patient the MDT have agreed have resectable lesions suspicious for pancreatic malignancy and going to surgery.

Benign Cohort

- Referral for endoscopic cystogastrostomy for complicated acute pancreatitis characterised by peripancreatic fluid collections and pseudocysts in development or matured (non-resolving and requiring further intervention).

OR

* Referral for cholecystectomy for cholocystitis/chololethiasis. OR
* Patient planned to have endoscopy investigation for dyspepsia (normal control subgroup).

Exclusion Criteria:

General

* Inability to provide written informed consent
* Other known malignant condition, either active or in complete remission ≤5 years
* HIV, hepatitis C, or any other known communicable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited into 3 groups. A group of pancreatic cancer patients will be selected from those diagnosed with localised pancreatic cancer, including both those undergoing successful resection, and those undergoing biopsy only (localised, but radiologically inoperable) or where resection was attempted.
  A control group will be formed from age- and gender-matched patients receiving hepatobiliary surgery or endoscopic intervention (ERCP, PTCA, instrumentation of the biliary tree, endoscopic cystogastrostomy for pancreatic pseudocyst) for benign inflammatory conditions.
  A third group of patients will be derived from those with suspected pancreatic cancer who are undergoing follow-up for pancreatic cystic lesions. HUTH provides an EUS service that at this point investigates about 40 such cystic lesions annually with paracentesis and has a significant number of cystic lesions under close follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of the accuracy of protein markers (e.g., TF, AM) in detecting early stage pancreatic cancer by comparison of laboratory results from ELISA assays and platform technologies to patient clinical data. | During the recruitment phase.
  The ELISAs and platform technologies will provide measurements of the markers (e.g. TF, AM) concentrations in patient urine, serum and cystic fluid samples. This will then be immediately linked to information on the pancreatic cancer diagnosis where it is known (i.e. cancer and control groups) and, for patients with pancreatic cysts, linked to information obtained following diagnostic work-up (and over the follow-up period), to determine the accuracy of these markers in the potential early detection of pancreatic cancer within the Hull University Teaching Hospitals NHS Trust (HUTH) pancreatic cancer population.
  Patients with a known cancer diagnosis, compared to controls, will be used to determine whether a suitable cut-off for each assay can be found for accurate detection.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Maraveyas, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Castle Hill Hospital, Hull University Teaching Hospitals NHS Trust, Cottingham, Kingston Upon Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No